CLINICAL TRIAL: NCT03832738
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of JTE-451 Administered for 16 Weeks in Subjects With Moderate to Severe Plaque Psoriasis (IMPACT-PS)
Brief Title: Study to Evaluate the Efficacy and Safety of JTE-451 in Subjects With Moderate to Severe Plaque Psoriasis
Acronym: IMPACT-PS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AE451-G-18-004
Record Dates: First submitted 2019-02-05; First posted 2019-02-06 (Actual); Results first posted 2021-08-16 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Plaque Psoriasis; Psoriasis; Skin Diseases
Keywords: JTE-451; Psoriasis; Plaque psoriasis; IMPACT-PS
MeSH Terms: conditions — Psoriasis; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- JTE-451 Dose 1 (Experimental): JTE-451 Tablets Dose 1 daily for 16 weeks.
  Interventions: Drug: JTE-451 Tablets
- JTE-451 Dose 2 (Experimental): JTE-451 Tablets Dose 2 daily for 16 weeks.
  Interventions: Drug: JTE-451 Tablets
- Placebo (Placebo Comparator): Placebo Tablets daily for 16 weeks.
  Interventions: Drug: Placebo Tablets

INTERVENTIONS:
Drug: JTE-451 Tablets — Active drug tablets containing JTE-451
  Arms: JTE-451 Dose 1; JTE-451 Dose 2
Drug: Placebo Tablets — Placebo tablets matching in appearance to the active drug tablets
  Arms: Placebo

SUMMARY:
Study to evaluate the efficacy and safety of JTE-451 administered for 16 weeks in subjects with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Have had a history of moderate to severe plaque psoriasis for at least 6 months prior to Visit 1;
* Subjects with moderate to severe plaque psoriasis covering ≥10% body surface area (BSA), with a psoriasis area and severity index (PASI) ≥12 and static Physician's Global Assessment (sPGA) score ≥3 at Visit 1 and Visit 2

Exclusion Criteria:

* History of discontinuation of biologic therapies (including marketed and investigational drugs) directly targeting Interleukin (IL)-17A, IL-17A/F, IL-17 receptor A, IL-12/IL-23p40 or IL-23p19 due to lack of efficacy, according to the Investigator's judgment;
* Prior exposure to retinoid-related orphan receptor (ROR)-γ inhibitors;
* Presence of erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis or other skin conditions (e.g., clinically-significant eczema or severe acne) at Visit 1;
* History or presence of itch due to underlying conditions other than plaque psoriasis which cause or influence pruritus of the skin within 12 months prior to Visit 1.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (6):
  - Clinical Science Institute, Santa Monica, California
  - Advanced Dermatology and Skin Cancer Specialists, Temecula, California
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Central Sooner Research, Norman, Oklahoma
  - Rhode Island Hospital, Providence, Rhode Island
  - Health Concepts, Rapid City, South Dakota
- Canada (6):
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - SKiN Health, Cobourg, Ontario
  - Research Toronto, Toronto, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
- Poland (21):
  - Szpital Uniwersytecki nr 1 im. Dr. A. Jurasza w Bydgoszczy, Klinika Dermatologii, Chorob Prenoszonych Droga Plciowa, Bydgoszcz
  - Copernicus Podmiot Leczniczy Sp. z o.o., Oddzial Dermatologii, Gdansk
  - Prywatny Gabinet Dermatologiczny Elzbieta Klujszo, Kielce
  - Centrum Nowoczesnych Terapii "Dobry Lekarz" Spolka z orgraniczona odpowiedzialnoscia, Krakow
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska Spolka Komandytowo-Akeyjna, Lodz
  - ETG Lodz, Lodz
  - Dermoklinika - Centrum Medyczne s.c., M. Kierstan, J. Narbutt, A. Lesiak, Lodz
  - ETG Lublin, Lublin
  - Centrum Medyczne Grunwald, Poznan
  - Solumed Centrum Medyczne, Poznan
  - Kliniczny Szpital Wojewodzki nr 1 im. Fryderyka Chopina w Rzeszowie, Klinika Dermatologii, Rzeszów
  - ETG Siedlce, Siedlce
  - ETG Skierniewice, Skierniewice
  - Clinical Research Group Sp. z o.o., Warsaw
  - Dorota Bystrzanowska "High-Med" Przychodnia Specjalistyczna, Warsaw
  - Carpe Diem Centrum Medycyny Estetycznej, Warsaw
  - Royalderm Agnieszka Nawrocka, Warsaw
  - ETG Warszawa, Warsaw
  - CITYCLINIC Przychodnia Psychologiczno-Lekarska Matusiak Spolka Partnerska, Wroclaw
  - DERMMEDICA Sp. z o.o., Wroclaw
  - ETG Zamosc, Zamość

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Written informed consent was obtained prior to performing any study-related procedures. A copy of the informed consent was provided to each subject enrolled in this study. To qualify for the study, subjects were required to satisfy defined criteria.
Pre-assignment Details: Following informed consent signing, screening procedures to confirm eligibility were performed.
  1. Intent-to-Treat (ITT) Population - 152 subjects
  2. Safety Population - 151 subjects
  3. Pharmacokinetic (PK) Population - 101 subjects
Groups:
- JTE-451 200 mg Twice Daily: JTE-451 200 mg orally twice daily for 16 weeks (total daily dose - 400 mg)
- JTE-451 400 mg Twice Daily: JTE-451 400 mg orally twice daily for 16 weeks (total daily dose - 800 mg)
- Placebo Twice Daily: Placebo Tablets orally twice daily for 16 weeks
Period: Overall Study
Arm/Group | JTE-451 200 mg Twice Daily | JTE-451 400 mg Twice Daily | Placebo Twice Daily
Started | 51 | 50 | 51
Completed | 43 | 38 | 32
Not Completed | 8 | 12 | 19
Not completed — Withdrawal by Subject | 6 | 7 | 16
Not completed — Physician Decision | 0 | 1 | 2
Not completed — Adverse Event | 2 | 3 | 1
Not completed — Pregnancy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics results are reported for the Intent-to-Treat (ITT) population: 152 randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | JTE-451 200 mg Twice Daily | JTE-451 400 mg Twice Daily | Placebo Twice Daily | Total
Number analyzed (Participants) | 51 | 50 | 51 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 47 | 46 | 46 | 139
  >=65 years | 4 | 4 | 5 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 21 | 16 | 50
  Male | 38 | 29 | 35 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 51 | 49 | 50 | 150
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0
  White | 51 | 47 | 49 | 147
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 5 | 5 | 3 | 13
  United States | 2 | 7 | 6 | 15
  Poland | 44 | 38 | 42 | 124
Prior exposure to biologics therapy [Count of Participants; unit: Participants]
  Had prior biologics therapy | 11 | 15 | 13 | 39
  No prior biologics therapy | 40 | 35 | 38 | 113
Body weight [Count of Participants; unit: Participants]
  Below 90 kg | 25 | 24 | 25 | 74
  90 kg or above | 26 | 26 | 26 | 78

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving a Minimum 75% Improvement From Baseline in the Psoriasis Area and Severity Index (PASI-75) at End-of-treatment (EOT)
Description: The psoriasis area and severity index (PASI) combines the assessment of the severity of lesions (scaling, redness and plaque thickness) and the area affected into a single score in the range of 0.0 (no disease) to 72.0 (maximal disease). The body is divided into four sections: (1) Head and neck; (2) Upper limbs; (3) Trunk (including axillae and groin); and (4) Lower limbs (including buttocks).
  The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis.
  The PASI-75 response rate is defined as at least 75 percent (%) reduction in PASI score at EOT (up to 16 weeks) relative to Baseline.
Time Frame: End of Treatment (Up to 16 Weeks)
Population: Subjects in the ITT Population at the EOT. The EOT value is defined as the last assessment during the treatment period (from the first dose of study drug to the last dose of study drug).
Measure: Number; unit: % of subjects achieving PASI-75
Arm/Group | JTE-451 200 mg Twice Daily | JTE-451 400 mg Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 51 | 50 | 51
% of subjects achieving PASI-75 | 11.8 | 22.0 | 7.8
Statistical Analysis 1: Comparison: JTE-451 200 mg Twice Daily vs Placebo Twice Daily; Test type: Superiority; p = 0.558, Cochran-Mantel-Haenszel — p-value was estimated based on Cochran-Mantel-Haenszel test stratified by prior exposure to biologic therapy (Yes/No) and body weight (<90 kg/≥90 kg); Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.39 to 5.80]
Statistical Analysis 2: Comparison: JTE-451 400 mg Twice Daily vs Placebo Twice Daily; Test type: Superiority; p = 0.035, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.74, 95% CI 2-sided [1.07 to 13.10]

2. Secondary Outcome: Percentage of Subjects Achieving a Minimum 50% Improvement From Baseline in the Psoriasis Area and Severity Index (PASI-50) at EOT
Description: The PASI combines the assessment of the severity of lesions (scaling, redness and plaque thickness) and the area affected into a single score in the range of 0.0 (no disease) to 72.0 (maximal disease). The body is divided into four sections: (1) Head and neck; (2) Upper limbs; (3) Trunk (including axillae and groin); and (4) Lower limbs (including buttocks).
  The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis.
  The PASI-50 response rate is defined as at least 50 percent (%) reduction in PASI score at EOT (up to 16 weeks) relative to Baseline.
Time Frame: End of Treatment (Up to 16 Weeks)
Population: as for outcome 1
Measure: Number; unit: % of subjects achieving PASI-50
Arm/Group | JTE-451 200 mg Twice Daily | JTE-451 400 mg Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 51 | 50 | 51
% of subjects achieving PASI-50 | 33.3 | 42.0 | 17.6
Statistical Analysis 1: Comparison: JTE-451 200 mg Twice Daily vs Placebo Twice Daily; Test type: Superiority; p = 0.086, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.26, 95% CI 2-sided [0.89 to 5.75]
Statistical Analysis 2: Comparison: JTE-451 400 mg Twice Daily vs Placebo Twice Daily; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.76, 95% CI 2-sided [1.45 to 9.75]

3. Secondary Outcome: Percentage of Subjects Achieving a Minimum 90% Improvement From Baseline in the Psoriasis Area and Severity Index (PASI-90) at EOT
Description: The PASI combines the assessment of the severity of lesions (scaling, redness and plaque thickness) and the area affected into a single score in the range of 0.0 (no disease) to 72.0 (maximal disease). The body is divided into four sections: (1) Head and neck; (2) Upper limbs; (3) Trunk (including axillae and groin); and (4) Lower limbs (including buttocks).
  The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis.
  The PASI-90 response rate is defined as at least 90 percent (%) reduction in PASI score at EOT (up to 16 weeks) relative to Baseline.
Time Frame: End of Treatment (Up to 16 Weeks)
Population: as for outcome 1
Measure: Number; unit: % of subjects achieving PASI-90
Arm/Group | JTE-451 200 mg Twice Daily | JTE-451 400 mg Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 51 | 50 | 51
% of subjects achieving PASI-90 | 2.0 | 6.0 | 2.0
Statistical Analysis 1: Comparison: JTE-451 200 mg Twice Daily vs Placebo Twice Daily; Test type: Superiority; p > 0.999, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1, 95% CI 2-sided [0.06 to 17.25]
Statistical Analysis 2: Comparison: JTE-451 400 mg Twice Daily vs Placebo Twice Daily; Test type: Superiority; p = 0.244, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.86, 95% CI 2-sided [0.36 to 41.20]

4. Secondary Outcome: Percent Change From Baseline in Psoriasis Area and Severity Index (PASI) Score at EOT
Description: The PASI combines the assessment of the severity of lesions (scaling, redness and plaque thickness) and the area affected into a single score in the range of 0.0 (no disease) to 72.0 (maximal disease). The body is divided into four sections: (1) Head and neck; (2) Upper limbs; (3) Trunk (including axillae and groin); and (4) Lower limbs (including buttocks).
  The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis.
  Percent change from baseline to EOT (up to 16 weeks) in PASI score was calculated by taking the PASI score at EOT and subtracting the baseline PASI score, then dividing by the baseline PASI score and multiplying by 100.
Time Frame: End of Treatment (Up to 16 Weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change in PASI Score
Arm/Group | JTE-451 200 mg Twice Daily | JTE-451 400 mg Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 51 | 50 | 48
% change in PASI Score | -30.33 (40.971) | -37.89 (37.896) | -17.53 (34.701)

5. Secondary Outcome: Percentage of Subjects Who Achieved Static Physician's Global Assessment (sPGA) Score of 0 or 1 at EOT
Description: The sPGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the redness, thickness and scaling across all psoriatic lesions. Average redness, thickness and scaling are scored separately over the whole body according to a 5-point severity scale (0 [no symptoms] to 4 [severe symptoms]). The total score is calculated as average of the 3 severity (redness, thickness and scaling) scores and rounded to the nearest whole number score to determine the sPGA score (0=cleared; 1=minimal; 2=mild; 3=moderate; and 4=severe).
  For this outcome measure, at EOT (up to 16 weeks), a score of 0 means no symptoms of psoriasis and a score of 1 means minimal symptoms of psoriasis.
Time Frame: End of Treatment (Up to 16 Weeks)
Population: as for outcome 1
Measure: Number; unit: % of subjects achieving sPGA 0 or 1
Arm/Group | JTE-451 200 mg Twice Daily | JTE-451 400 mg Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 51 | 50 | 51
% of subjects achieving sPGA 0 or 1 | 25.5 | 28.0 | 5.9
Statistical Analysis 1: Comparison: JTE-451 200 mg Twice Daily vs Placebo Twice Daily; Test type: Superiority; p = 0.009, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 5.21, 95% CI 2-sided [1.38 to 19.62]
Statistical Analysis 2: Comparison: JTE-451 400 mg Twice Daily vs Placebo Twice Daily; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 7.35, 95% CI 2-sided [1.86 to 29.08]

6. Secondary Outcome: Change From Baseline in Static Physician's Global Assessment (sPGA) Score at EOT
Description: The sPGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the redness, thickness and scaling across all psoriatic lesions. Average redness, thickness and scaling are scored separately over the whole body according to a 5-point severity scale (0 [no symptoms] to 4 [severe symptoms]). The total score is calculated as average of the 3 severity (redness, thickness and scaling) scores and rounded to the nearest whole number score to determine the sPGA score (0=cleared; 1=minimal; 2=mild; 3=moderate; and 4=severe).
  Change from baseline to EOT (up to 16 weeks) in sPGA score was calculated by taking the sPGA score at EOT and subtracting the baseline sPGA score.
Time Frame: End of Treatment (Up to 16 Weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JTE-451 200 mg Twice Daily | JTE-451 400 mg Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 51 | 50 | 48
score on a scale | -0.96 (0.848) | -1.02 (0.869) | -0.54 (0.713)

7. Secondary Outcome: Percent Change From Baseline in Psoriasis Body Surface Area (BSA) at EOT
Description: The total body surface area (BSA) affected by plaque-type psoriasis was obtained from the percentages of areas affected, including head, trunk, upper limbs and lower limbs. Each reported percentage was multiplied by its respective body region corresponding factor (head=0.1, upper limbs=0.2, trunk=0.3, lower limbs=0.4) and the resulting 4 values were added up to obtain the total psoriasis BSA (Range: 0 to 100).
  BSA (%)=0.1Sh+0.2Su+0.3St+0.4Sl, where S=body region surface area with psoriasis: h=head; u=upper limbs; t=trunk; l=lower limbs.
  Percent change from baseline to EOT (up to 16 weeks) in BSA was calculated by taking the EOT BSA and subtracting the baseline BSA, then dividing by the baseline BSA and multiplying by 100.
  A negative change from baseline at EOT indicates a reduction in the Psoriasis BSA compared to the baseline.
Time Frame: End of Treatment (Up to 16 Weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % Change in Psoriasis BSA
Arm/Group | JTE-451 200 mg Twice Daily | JTE-451 400 mg Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 51 | 50 | 48
% Change in Psoriasis BSA | -18.67 (39.582) | -19.03 (48.696) | -5.74 (38.707)

8. Secondary Outcome: Change From Baseline in the Skindex-16 Overall Score at EOT
Description: Skindex-16 questionnaire contains 16 questions related to quality of life in subjects with skin disease. It consists of a short 16-item assessment completed by the subject, with each item rated on a 7-point Likert scale (0=never bothered to 6=always bothered). Each raw score is multiplied by 16.667 to transform all responses to a linear scale from 0 (no effect) to 100 (effect experienced all the time). Responses to the Skindex-16 are categorized into 3 subscales: symptom, emotional & functional; their respective scores are expressed in a linear scale from 0 to 100. Overall scale score is an average of 16 items expressed in a linear scale from 0 to 100.
  Change from baseline to EOT (up to 16 weeks) in the Skindex-16 Overall Score was calculated by taking the EOT Skindex-16 Overall Score and subtracting the baseline Skindex-16 Overall Score.
  A negative change from baseline at EOT indicates an improvement in the subject's condition compared to the baseline.
Time Frame: End of Treatment (Up to 16 Weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JTE-451 200 mg Twice Daily | JTE-451 400 mg Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 51 | 50 | 48
score on a scale | -10.029 (23.2635) | -10.896 (26.7910) | -3.386 (20.8617)

9. Secondary Outcome: Change From Baseline in the Skindex-16 Symptom Scale Scores at EOT
Description: Skindex-16 questionnaire contains 16 questions related to quality of life in subjects with skin disease. It consists of a short 16-item assessment completed by the subject, with each item rated on a 7-point Likert scale (0=never bothered to 6=always bothered). Each raw score is multiplied by 16.667 to transform all responses to a linear scale from 0 (no effect) to 100 (effect experienced all the time). Responses to the Skindex-16 are categorized into 3 subscales: symptom, emotional & functional; their respective scores are expressed in a linear scale from 0 to 100. Symptoms scale score is an average of items 1 to 4 expressed in a linear scale from 0 to 100.
  Change from baseline to EOT (up to 16 weeks) in the Skindex-16 Symptoms Scale Score was calculated by taking the EOT Skindex-16 Symptoms Scale Score and subtracting the baseline Skindex-16 Symptoms Scale Score.
  A negative change from baseline at EOT indicates an improvement in the subject's condition compared to the baseline.
Time Frame: End of Treatment (Up to 16 Weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JTE-451 200 mg Twice Daily | JTE-451 400 mg Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 51 | 50 | 48
score on a scale | -8.905 (34.2989) | -11.500 (31.5148) | -2.170 (26.0563)

10. Secondary Outcome: Change From Baseline in the Skindex-16 Emotions Scale Scores at EOT
Description: Skindex-16 questionnaire contains 16 questions related to quality of life in subjects with skin disease. It consists of a short 16-item assessment completed by the subject, with each item rated on a 7-point Likert scale (0=never bothered to 6=always bothered). Each raw score is multiplied by 16.667 to transform all responses to a linear scale from 0 (no effect) to 100 (effect experienced all the time). Responses to the Skindex-16 are categorized into 3 subscales: symptom, emotional & functional; their respective scores are expressed in a linear scale from 0 to 100. Emotions scale score is an average of items 5 to 11 expressed in a linear scale from 0 to 100.
  Change from baseline to EOT (up to 16 weeks) in the Skindex-16 Emotions Scale Score was calculated by taking the EOT Skindex-16 Emotions Scale Score and subtracting the baseline Skindex-16 Emotions Scale Score.
  A negative change from baseline at EOT indicates an improvement in the subject's condition compared to the baseline.
Time Frame: End of Treatment (Up to 16 Weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JTE-451 200 mg Twice Daily | JTE-451 400 mg Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 51 | 50 | 48
score on a scale | -10.411 (21.8268) | -13.143 (28.4467) | -5.953 (22.6358)

11. Secondary Outcome: Change From Baseline in the Skindex-16 Functioning Scale Scores at EOT
Description: Skindex-16 questionnaire contains 16 questions related to quality of life in subjects with skin disease. It consists of a short 16-item assessment completed by the subject, with each item rated on a 7-point Likert scale (0=never bothered to 6=always bothered). Each raw score is multiplied by 16.667 to transform all responses to a linear scale from 0 (no effect) to 100 (effect experienced all the time). Responses are categorized into 3 subscales: symptom, emotional & functional; their respective scores are expressed in a linear scale from 0 to 100. Functioning scale score is an average of items 12 to 16 expressed in a linear scale from 0 to 100.
  Change from baseline to EOT (up to 16 weeks) in the Skindex-16 Functioning Scale Score was calculated by taking the EOT Skindex-16 Functioning Scale Score and subtracting the baseline Skindex-16 Functioning Scale Score.
  A negative change from baseline at EOT indicates an improvement in the subject's condition compared to the baseline.
Time Frame: End of Treatment (Up to 16 Weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JTE-451 200 mg Twice Daily | JTE-451 400 mg Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 51 | 50 | 48
score on a scale | -10.392 (23.5294) | -7.267 (27.6823) | -0.764 (20.1090)

12. Secondary Outcome: Change From Baseline in Itch Numeric Rating Scale (NRS) at EOT
Description: The Itch NRS is a validated, self-reported, instrument for measurement of itch intensity and subjects were asked to rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable); higher scores indicated greater itch intensity. The Itch NRS scores were recorded by the subject using the e-diary once daily from screening through the last visit.
  Change from baseline to EOT (up to 16 weeks) in the Itch NRS Score was calculated by taking the Itch NRS Score (weekly average) at EOT and subtracting the baseline Itch NRS Score (weekly average).
Time Frame: End of Treatment (Up to 16 Weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JTE-451 200 mg Twice Daily | JTE-451 400 mg Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 51 | 50 | 48
score on a scale | -1.302 (2.8165) | -1.537 (3.2634) | -0.547 (2.4239)

13. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse Events
Description: Subjects in the Safety Population (151, randomized subjects who received at least one dose of study drug).
  The treatment-emergent adverse event (TEAE) is defined as one of the following:
  1. An adverse event (AE) that occurred during the treatment period or the follow-up period. In the process of collecting the onset dates of AEs, an AE that occurs after the initiation of trial medication on Day 1 (the first day of the treatment period) should be treated as a TEAE. All AEs occurring on the day of first dose will be considered as TEAE if the time of AE occurrence relative to the dosing is unknown.
  2. An AE present prior to the treatment period that worsened in severity during the treatment period or the follow-up period.
  3. Any events that are present prior to the treatment period and have recovered, but recurred during the treatment period or the follow-up period should be considered as new TEAEs.
Time Frame: Follow-up (Up to 20 Weeks)
Population: Safety Population (151, randomized subjects who received at least one dose of study drug).
Measure: Count of Participants; unit: Participants
Arm/Group | JTE-451 200 mg Twice Daily | JTE-451 400 mg Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 51 | 50 | 50
Participants
  Number of subjects with TEAEs | 27 | 28 | 25
  Number of subjects with no TEAEs | 24 | 22 | 25

14. Secondary Outcome: JTE-451 Trough Plasma Concentrations at Week 16
Description: Trough plasma concentration is the measured concentration at the end of a dosing interval at steady state (taken directly before next administration). Blood samples were collected at specific timepoints to measure trough plasma concentration of JTE-451 in the pharmacokinetic (PK) population.
Time Frame: Week 16
Population: Subjects (75 subjects) in the PK population at Week 16 with available trough plasma concentrations of JTE-451 (subjects who received at least one dose of JTE-451 and have at least one usable JTE-451 plasma concentration measurement at Week 16).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | JTE-451 200 mg Twice Daily | JTE-451 400 mg Twice Daily
Number analyzed (Participants) | 42 | 33
ng/mL | 575 (704) | 1210 (1660)

ADVERSE EVENTS:
Time Frame: Up to 20 Weeks
Description: Subjects in the Safety Population (151, randomized subjects who received at least one dose of study drug).
Arm/Group | JTE-451 200 mg Twice Daily | JTE-451 400 mg Twice Daily | Placebo Twice Daily
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/51 | 2/50 | 1/50
Other Adverse Events (participants affected / at risk) | 20/51 | 22/50 | 17/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JTE-451 200 mg Twice Daily (N=51) | JTE-451 400 mg Twice Daily (N=50) | Placebo Twice Daily (N=50)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Breast Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JTE-451 200 mg Twice Daily (N=51) | JTE-451 400 mg Twice Daily (N=50) | Placebo Twice Daily (N=50)
Hypertension (Vascular disorders) | 2 (3) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 3 (3) | 1 (1)
Blood Glucose Increased (Investigations) | 2 (2) | 1 (1) | 2 (2)
Gamma-Glutamyltransferase Increased (Investigations) | 2 (2) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 4 (8) | 1 (1) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 4 (4) | 2 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (13) | 19 (30) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (4) | 2 (2) | 5 (5)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 3 (3) | 4 (4)
Urinary Tract Infection (Infections and infestations) | 3 (4) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT03832738/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT03832738/SAP_001.pdf